CLINICAL TRIAL: NCT03752424
Title: Topical Silver Nanoparticles for Microbial Activity
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed A. H. Abdellatif (Other)
Responsible Party: Sponsor-Investigator, Ahmed A. H. Abdellatif, Assistant Professor of Pharmaceutics, Faculty of Pharmacy, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharSilver
Record Dates: First submitted 2018-11-10; First posted 2018-11-26 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Foot Infection Fungal; Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — colloidal silver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver nanoparticles group (Active Comparator): A group of volunteers infected with Tinea pedis, Capitis and Versicolor received Topical silver nanoparticles in different dosage forms.
  Interventions: Drug: Silver nanoparticles
- Topical approved anti-microbial gel (Placebo Comparator): A group of volunteers infected with Tinea pedis, Capitis and Versicolor received placebo cream.
  Interventions: Drug: Topical approved anti-microbial gel

INTERVENTIONS:
Drug: Silver nanoparticles — The active group will receive silver nanoparticles in different dosage forms as an anti-microbial drug.
  Other Names: Topical jel
  Arms: Silver nanoparticles group
Drug: Topical approved anti-microbial gel — The placebo group will receive topical FDA approved anti-microbial jel in different dosage forms as control drug.
  Other Names: Topical anti-microbial gel
  Arms: Topical approved anti-microbial gel

SUMMARY:
Silver nanoparticles are one of most nanoparticles use nowadays in the research area because it has specific physical and chemical properties, in medical fields silver nanoparticles can involve in diagnostic and treatment processes. Silver nanoparticles have antibacterial, antiviral, antifungal, antiangiogenic, antioxidant, cosmetics, antitumor, anti-inflammatory, the drug carrier, imaging, water treatment, and biosensing effects. Silver nanoparticles prepared with reducing agent tri-sodium citrate then incorporated in a topical cream to obtain a significant inhibition of the bacterial strains, inhibition of growth of bacterial strains in the face or other parts in the bodies.

DETAILED DESCRIPTION:
1. Preparation of vanishing cream Vanishing cream is an emulsion base which is oil in water, the oil phase gives the cream shine and pearl look because of stearic acid in the oil. To form an emulsion, the alkali will react with stearic acid to form stearate soap. Then mix sodium hydroxide (NaOH) with potassium hydroxide (KOH) to give cream hard and soft properties.
2. Preparation of cream containing silver nanoparticles Silver nanoparticles will be produced by using the reduction reaction method. The reaction involves heating silver nitrate at a high temperature with adding a reducing agent, the particles will produce as silver nanoparticles in liquid form.
3. Characterization of the Vanishing cream containing drug:

   3.1. Drug content: The amount of drug in cream will be determined by taking 100 mg of the cream formulation and dissolve it in 10 mL of methanol after that it will be filtrated. In addition, it will be analyzed the content of drug spectrophotometrically using (UV-VIS) at specific λmax.

   3.2. Irritation to skin: In this test, the cream formulation will be applied to four healthy volunteers which they should not have any sensitivity to the drug. They will inform about the nature of the formulation and obtain a written approval from them about the irritation effect of the formulated cream.
4. Anti-microbial studies:

The antifungal action for formula will be studied using different 6 groups volunteers The inhibition microbial activity for all formulae were compared with known standard antimicrobial drugs.

ELIGIBILITY:
Inclusion Criteria:

* It is important to follow up and collect data, preferably for six months for the local and systemic activity of silver nanoparticles, to establish whether the infection recurrent or not.

Exclusion Criteria:

* Larger numbers of participants having a different kind of skin infection are needed to test efficiency drug in order to produce more reliable data.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-13 (Estimated); Primary Completion 2020-01-12 (Estimated); Study Completion 2021-01-11 (Estimated)

PRIMARY OUTCOMES:
The antimicrobial activity of silver nanoparticles in the two groups of control and an infected patient will be determined. Each group will be of 6 volunteers, each one will be controlled for the CTCAE. | Six months
  The formulated silver nanoparticles are expected to be with anti-microbial after applying activity with infected patients even systemically or topically. The nanoparticles will be examined on two groups of patients (control group, and patient with fungal or microbial infections). Moreover, the obtained silver nanoparticles are expected to highly internalized and disease targeted. The results will be compared with control groups to prove the anti-microbial Activity. The progress of treating the patient will be noticed by completely disappear of fungal infection.

SECONDARY OUTCOMES:
Stable topical anti-microbial silver nanoparticles | three months
  Stability test will be studied for dosage forms. The test will carried out by standing the products on shelf life for three months. The stability test will be recorded using high performance liquid chromatography each thee days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AH Abdellatif, PhD, Principal Investigator — Qassim University
Locations (1):
- Buraidah Clinic, Buraidah, Al Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The authors could not decide until now a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Gunasekaran T, Nigusse T, Dhanaraju MD. Silver nanoparticles as real topical bullets for wound healing. J Am Coll Clin Wound Spec. 2012 Jun 4;3(4):82-96. doi: 10.1016/j.jcws.2012.05.001. eCollection 2011 Dec. PMID 24527370